CLINICAL TRIAL: NCT06449716
Title: A Tailored Intervention to Prevent Age-Related Declines in Muscle Power and Functional Ability
Brief Title: Tailored Versus Traditional Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Christophe Delecluse, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S68434
Record Dates: First submitted 2024-03-05; First posted 2024-06-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Exercise Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized resistance exercise program (Experimental): Individualized exercise dose. Individuals with a velocity deficit only perform low-load exercises. Individuals with a force deficit only perform high-load exercises.
  Interventions: Other: 12-week progressive power-oriented resistance exercise program
- Non-individualized resistance exercise program (Active Comparator): Non-individualized exercise dose. All individuals perform a combination of low-load and high-load resistance exercises, regardless of their deficit.
  Interventions: Other: 12-week progressive power-oriented resistance exercise program

INTERVENTIONS:
Other: 12-week progressive power-oriented resistance exercise program — 2x/week, 35-45 min sessions, on leg press machine

SUMMARY:
Preserving functional ability is crucial for healthy aging. Unfortunately, age-related decreases in muscle power often lead to declines in functional ability. As power is the product of force and velocity, decreases in power can originate from changes in muscle force, contraction velocity, or both, varying between individuals. The primary method to prevent functional disability is power-based resistance training. Although training interventions are effective for most older adults, they do not induce substantial improvements in a subset of the population. These inconsistent outcomes may arise from neglecting the observed differences in the force-velocity (F-v) profiles between individuals. Therefore, this study provides a novel approach to resistance exercise, in which exercise dose is tailored according to the individual's F-v profile. The effectiveness of the tailored method will be assessed in a randomized control trial, comparing the effects of an individualized and a non-individualized 12-week training intervention on muscle power parameters and functional ability.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults
* 65-80 years old

Exclusion Criteria:

* Systematic engagement in resistance exercise during the past year
* Unstable cardiovascular disease, neuromuscular disease, acute infection or fever
* Recent surgery
* Lower-extremity injuries
* Low levels of functional ability (i.e., SPPB score ≤ 9)
* Cognitive malfunctioning (i.e., Mini-Mental State Examination < 24)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-12-04 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
Maximal force (F0) | Change from baseline in maximal force at 12 weeks
  Unilateral (dominant leg) maximal force production (N) on the pneumatic leg press device (Leg Press Air 400, Keiser, USA).
  The test protocol consists of 2 sets of 1 repetition with increasing loads (5-10 kg increments), starting at 20% of body mass. When the participants fail to lift a certain load, the load will be decreased by 2.5-5 kg until their one repetition maximum (1-RM) is reached. The duration of the recovery time between sets will be based on the mean velocity in the preceding repetition, with longer rest periods after high-load, low-velocity attempts. Mean velocity of the best trial per load is used to estimate the individual F-v relationship through a linear equation. This F-v relationship will be used to examine the exercise-induced changes in maximal force.
Maximal velocity (V0) | Change from baseline in maximal velocity at 12 weeks
  Unilateral (dominant leg) maximal velocity production (m/s) on the pneumatic leg press device (Leg Press Air 400, Keiser, USA).
  The test protocol consists of 2 sets of 1 repetition with increasing loads (5-10 kg increments), starting at 20% of body mass. When the participants fail to lift a certain load, the load will be decreased by 2.5-5 kg until their one repetition maximum (1-RM) is reached. The duration of the recovery time between sets will be based on the mean velocity in the preceding repetition, with longer rest periods after high-load, low-velocity attempts. Mean velocity of the best trial per load is used to estimate the individual F-v relationship through a linear equation. This F-v relationship will be used to examine the exercise-induced changes in maximal velocity.
Force-velocity slope | Change from baseline in F-v slope at 12 weeks
  Unilateral (dominant leg) force-velocity (F-v) slope on the pneumatic leg press device (Leg Press Air 400, Keiser, USA). F-v slope = force (N) as a function of velocity (m/s).
  The test protocol consists of 2 sets of 1 repetition with increasing loads (5-10 kg increments), starting at 20% of body mass. When the participants fail to lift a certain load, the load will be decreased by 2.5-5 kg until their one repetition maximum (1-RM) is reached. The duration of the recovery time between sets will be based on the mean velocity in the preceding repetition, with longer rest periods after high-load, low-velocity attempts. Mean velocity of the best trial per load is used to estimate the individual F-v relationship through a linear equation. This F-v relationship will be used to examine the exercise-induced changes in slope.
Maximal power (P0) | Change from baseline in maximal power at 12 weeks
  Unilateral (dominant leg) maximal power production (Watt) on the pneumatic leg press device (Leg Press Air 400, Keiser, USA).
  The test protocol consists of 2 sets of 1 repetition with increasing loads (5-10 kg increments), starting at 20% of body mass. When the participants fail to lift a certain load, the load will be decreased by 2.5-5 kg until their one repetition maximum (1-RM) is reached. The duration of the recovery time between sets will be based on the mean velocity in the preceding repetition, with longer rest periods after high-load, low-velocity attempts. Mean velocity of the best trial per load is used to estimate the individual F-v relationship through a linear equation. This F-v relationship will be used to examine the exercise-induced changes in maximal power.
Force at maximal power | Change from baseline in force at maximal power at 12 weeks
  Unilateral (dominant leg) force at maximal power production (N) on the pneumatic leg press device (Leg Press Air 400, Keiser, USA).
  The test protocol consists of 2 sets of 1 repetition with increasing loads (5-10 kg increments), starting at 20% of body mass. When the participants fail to lift a certain load, the load will be decreased by 2.5-5 kg until their one repetition maximum (1-RM) is reached. The duration of the recovery time between sets will be based on the mean velocity in the preceding repetition, with longer rest periods after high-load, low-velocity attempts. Mean velocity of the best trial per load is used to estimate the individual F-v relationship through a linear equation. This F-v relationship will be used to examine the exercise-induced changes in force at maximal power.
Velocity at maximal power | Change from baseline in velocity at maximal power at 12 weeks
  Unilateral (dominant leg) velocity at maximal power production (m/s) on the pneumatic leg press device (Leg Press Air 400, Keiser, USA).
  The test protocol consists of 2 sets of 1 repetition with increasing loads (5-10 kg increments), starting at 20% of body mass. When the participants fail to lift a certain load, the load will be decreased by 2.5-5 kg until their one repetition maximum (1-RM) is reached. The duration of the recovery time between sets will be based on the mean velocity in the preceding repetition, with longer rest periods after high-load, low-velocity attempts. Mean velocity of the best trial per load is used to estimate the individual F-v relationship through a linear equation. This F-v relationship will be used to examine the exercise-induced changes in velocity at maximal power.

SECONDARY OUTCOMES:
Exercise adherence | Total adherence over 12-week period
  Number of sessions attended as a percentage of total sessions planned
Short Physical Performance Battery (SPPB) score | Change from baseline in SPPB test score at 12 weeks
  Total score on the SPPB (min 0, max 12, higher scores indicate better performance)
Gait speed | Change from baseline in gait speed at 12 weeks
  The average speed (m/s) to walk 10m as fast as possible
Countermovement jump height | Change from baseline in countermovement jump height at 12 weeks
  The jump height (cm) in a countermovement jump
Timed up and go | Change from baseline in timed up and go time at 12 weeks
  The time (s) needed to stand up from a chair, walk 3 m, turn, walk back and sit down again (as fast as possible)
5-repetition sit-to-stand time | Change from baseline in sit-to-stand performance at 12 weeks
  The time (s) needed to perform 5 sit-to-stand transitions
5-repetition sit-to-stand power | Change from baseline in sit-to-stand performance at 12 weeks
  The power (watt) needed to perform 5 sit-to-stand transitions
Stair ascent time | Change from baseline in stair climbing performance at 12 weeks
  The time (s) needed to ascend a flight of stairs
Stair ascent power | Change from baseline in stair climbing performance at 12 weeks
  The power (Watt) needed to ascend a flight of stairs

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven - Department of Movement Sciences, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No